CLINICAL TRIAL: NCT05563025
Title: Comparison of Time and Cost Efficiency in Arthroscopic Shoulder Surgery Under Regional Anesthesia vs General Anesthesia
Acronym: vs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Other Study IDs: SamsunU_Art_Should_cost
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Anesthesia
Keywords: Cost; Regional Anesthesia; Shoulder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General: Arthroscopic Shoulder Surgery under General Anesthesia
- Regional: Arthroscopic Shoulder Surgery under Regional Anesthesia

SUMMARY:
Arthroscopic Shoulder surgery can be done not only under general anesthesia but also regional technics. In this study we aimed to compare the cost and time effectiveness of regional anesthesia and general anesthesia.

DETAILED DESCRIPTION:
In our routine practice, ultrasound guided brachial plexus blocks or general anesthesia can be used during shoulder surgery. This retrospective study is designed to investigate the data of the patients who underwent arthroscopic shoulder between 01.09.2021-01.09.2022 at Samsun University Education and Research Hospital. As well as patients' demographic data, presence of additional diseases, operation indications, duration of surgery, intraoperative medical agents that are used, duration of hospital stay will be collected from patients files.Fees for materials used for general anesthesia and regional anesthesia will be determined. A fixed cost will be determined for the use of the operating room, including the salaries of the healthcare workers. After final calculation of both of the group costs statistical analysis will be made.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) 1-2-3
* Arthroscopic Shoulder Surgery

Exclusion Criteria:

* Emergency surgery
* ASA -4

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients between age 18 and 80 of ASA status 1,2,3 who underwent Arthroscopic Shoulder Surgery under General or Regional Anesthesia between 01.09.2021 and 01.09.2022.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-12-16 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Cost of Regional Anesthesia and General Anesthesia | 1 year
  Calculation of peroperative costs of patients undergoing arthroscopic shoulder surgery under general or regional anesthesia. excluding surgical materials

SECONDARY OUTCOMES:
Time | 1 year
  Measuring the operation room usage under general or regional anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Tulgar, Study Chair — Samsun University
Locations (1):
- Samsun University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tapar H, Suren M, Kaya Z, Arıcı S, Karaman S, Kahveci M. Üst Ekstremite Periferik Blok Anestezisi Ve Komplikasyonları. Journal of Contemporary Medicine 2012;2(3):195-200.
- [Background] Hewson DW, Oldman M, Bedforth NM. Regional anaesthesia for shoulder surgery. BJA Educ. 2019 Apr;19(4):98-104. doi: 10.1016/j.bjae.2018.12.004. Epub 2019 Feb 6. No abstract available. PMID 33456877
- [Background] Komann M, Avian A, Dreiling J, Gerbershagen H, Volk T, Weinmann C, Meissner W. Association of Perioperative Regional Analgesia with Postoperative Patient-Reported Pain Outcomes and Opioid Requirements: Comparing 22 Different Surgical Groups in 23,911 Patients from the QUIPS Registry. J Clin Med. 2021 May 19;10(10):2194. doi: 10.3390/jcm10102194. PMID 34069496
- [Background] Gonano C, Kettner SC, Ernstbrunner M, Schebesta K, Chiari A, Marhofer P. Comparison of economical aspects of interscalene brachial plexus blockade and general anaesthesia for arthroscopic shoulder surgery. Br J Anaesth. 2009 Sep;103(3):428-33. doi: 10.1093/bja/aep173. Epub 2009 Jul 8. PMID 19586958